CLINICAL TRIAL: NCT04497519
Title: Local Tolerability and Pharmacokinetic Evaluation of Cyclops Dry Powder Hydroxychloroquine Inhalation in Healthy Volunteers; a Pilot Study
Brief Title: Local Tolerability and Pharmacokinetic Evaluation of Cyclops Dry Powder Hydroxychloroquine Inhalation in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Onno Akkerman, Principal Investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARRIED-01
Record Dates: First submitted 2020-07-27; First posted 2020-08-04 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Healthy volunteers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: inhaled hydroxychloroquine — ascending dose of iHCQ

SUMMARY:
Rationale:

This protocol describes a study on the local tolerability of dry powder hydroxychloroquine using the Cyclops in healthy volunteers.

Objective:

* Primary objective is to assess the local tolerability of dry powder hydroxychloroquine sulphate via the Cyclops at different dosages.
* Secondary objective is to investigate systemic pharmacokinetic parameters of dry powder hydroxychloroquine sulphate via the Cyclops at different dosages.

Study design: single center, ascending dose study Study population: twelve healthy volunteers

Main study parameters/endpoints:

The local tolerability of the inhalation of dry powder hydroxychloroquine sulphate (5, 10 and 20 mg) defined by a lung function deterioration (a drop of forced expiratory volume in 1 second (FEV1) of >15%), cough, or any other reported adverse event. Pharmacokinetic parameters will be derived from calculated actual inhaled dose (dose minus remainder in inhaler after inhalation) and in blood samples drawn pre-dose, at 0.5 and 2 and 3.5 hrs after inhalation. The inspiratory parameters during the inhalation maneuver are critical to explore predictors for drug exposure. The following parameters will be measured/calculated: dPmax (maximum pressure drop), Vi (inhaled volume), Ti (total inhalation time), PIF (peak inspiratory flow rate), MIF (mean inspiratory flow rate) and the FIR (average flow increase rate between 20% and 80% of PIF).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The participants included are healthy volunteers. They will receive three different doses of hydroxychloroquine sulphate using the dry powder inhaler (DPI) with (at least) seven days in between doses. Before using the dry powder inhaler (DPI), they will receive instructions and their inspiratory flow will be tested. To investigate local tolerability, lung function tests will be performed, and the occurrence of adverse events will be scored. Furthermore, before each test dose an indwelling cannula will be inserted and blood samples will be taken before and after each test dose. Four blood samples will be collected with each inhaled dose. Finally, five ECGs will be obtained to monitor for QT prolongation, one at the screenings visit, one at base-line and one after each inhalation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Age 18-65 years
* Obtained written informed consent

Exclusion Criteria:

1. Pregnancy or breastfeeding. Women in the fertility period and without using proper contraceptives will undergo a urine pregnancy test.
2. Contra-indication to (hydroxy)chloroquine or quinine (allergic reaction, prolonged QTc-interval (> 450 msec), long-QT syndrome (LQTS), retinopathy, epilepsia, myasthenia gravis, G6PD-deficiency).
3. Concurrent use of ciclosporin, digoxin, ritonavir, tamoxifen or tranylcypromine.
4. Concurrent use of high risk QTc prolongating drugs (amiodarone, erythromycin (daily dose > 1000 mg) or sotalol)16.
5. COVID-19 like symptoms, such as fever, couch, or sore throat; only by history taking.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Local tolerability | 35 minutes after inhalation
  Number of patients with a lung function deterioration (a drop of forced expiratory volume in 1 second (FEV1) of >15%.
Local tolerability | 95 minutes after inhalation
  Number of patients with a lung function deterioration (a drop of forced expiratory volume in 1 second (FEV1) of >15%.
Local tolerability | 5 hours
  Number of patients that report cough, or any other adverse event after inhalation.

SECONDARY OUTCOMES:
Pharmacokinetic parameter | 0,5 hour
  Calculated actual inhaled dose
Pharmacokinetic parameter | 3,5 hours
  Cmax
Pharmacokinetic parameter | 3,5 hours
  Tmax

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No